CLINICAL TRIAL: NCT01497093
Title: A Phase 1, Multicenter, Open Label, Dose-escalation Study to Determine the Maximum Tolerated Dose for the Combination of Pomalidomide (POM), Bortezomib (BTZ) and Low-Dose Dexamethasone (LDDEX) in Subjects With Relapsed or Refractory Multiple Myeloma (MM)
Brief Title: Study to Determine the Maximum Tolerated Dose for the Combination of Pomalidomide, Bortezomib and Low-Dose Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Multiple Myeloma Research Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-005
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; Relapsed Multiple Myeloma; Relapsed and Refractory Multiple Myeloma; Refractory Myeloma; Resistant Multiple Myeloma; Treatment-resistant Multiple Myeloma; Pomalidomide; Lenalidomide-resistant
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — pomalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pomalidomide/Bortezomib/Dexamethasone (Experimental): 1, 2, 3 or 4 mg of pomalidomide will be taken orally on Days 1-14 of a 21-day cycle along with 1 or 1.3 mg/m2 of bortezomib administered intravenously or subcutaneously on Days 1, 4, 8 and 11 of 21 days for cycles 1 -8 and on days 1, 8 of 21 days for cycle 9 and onward until disease progression, and dexamethasone 20 mg/day [≤ 75 years old] or 10 mg/day [> 75 years old] orally on days 1, 2, 4, 5, 8, 9, 11, 12 of 21 days for cycles 1-8 and on days 1, 2, 8, 9 of 21 days for cycles 9 and onward until disease progression
  Interventions: Drug: Pomalidomide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — Pomalidomide 1, 2, 3, or 4 mg will be taken orally on Days 1-14 of a 21-day cycle
  Other Names: CC-4047; Oral Pomalidomide
Drug: Bortezomib — Bortezomib 1 or 1.3 mg/m2 will be administered intravenously or subcutaneously on Days 1, 4, 8 and 11 of 21 days for cycles 1 -8 and on days 1, 8 of 21 days for cycle 9 and onward until disease progression
  Other Names: Velcade
Drug: Dexamethasone — Dexamethasone 20 mg/day [≤ 75 years old] or 10 mg/day [> 75 years old] will be taken orally on days 1, 2, 4, 5, 8, 9, 11, 12 of 21 days for cycles 1-8 and on days 1, 2, 8, 9 of 21 days for cycles 9 and onward until disease progression

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of pomalidomide in combination with bortezomib and low-dose dexamethasone in subjects with relapsed or refractory multiple myeloma

DETAILED DESCRIPTION:
A 3 + 3 design will be utilized to determine the MTD for POM + IV BTZ + LD-DEX combination treatment in a 21-day treatment cycle. DLT will be assessed to determine MTD during the first treatment cycle. Once the MTD is determined or the maximum planned dose (MPD) is reached without reaching MTD for POM + IV BTZ + LD-DEX, a cohort of 6 additional subjects will be treated at this MTD/MPD level to further confirm the safety and assess preliminary efficacy. An additional cohort of subjects will be enrolled to explore the safety for the combination of POM + BTZ + LD-DEX when using SQ BTZ. Subject in this cohort will receive POM + BTZ + LD-DEX at the MTD/MPD level per the MTD determination part of the study, except, the BTZ will be administered subcutaneously (SQ) instead of intravenously (IV). In, Protocol Amendment #4, the number of subject enrolled to be enrolled into the exploratory SQ BTZ cohort was increased from 6 to 12.

ELIGIBILITY:
Inclusion criteria:

1. Must be ≥ 18 years at the time of signing the informed consent form.
2. Subjects must have documented diagnosis of multiple myeloma and have measurable disease (serum M-protein ≥ 0.5 g/dL or urine M-protein ≥ 200 mg/24 hours).
3. Subjects must have had at least 1 but no greater than 4 prior anti-myeloma therapies.
4. Subjects must have received at least 2 consecutive cycles of prior treatment with lenalidomide and must be refractory to their last lenalidomide-containing regimen (either as a single agent or in combination).
5. Subjects must have received at least 2 consecutive cycles of prior treatment with a proteasome inhibitor-containing regimen, but must not be refractory to bortezomib (either as a single agent or in combination).
6. Subjects must have documented progression during or after their last anti-myeloma therapy.
7. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.

Exclusion criteria:

1. Subjects who are refractory to bortezomib either as single agent or in combination.
2. Subjects with peripheral neuropathy ≥ Grade 2
3. Subjects with non-secretory multiple myeloma
4. Subjects with any of the following laboratory abnormalities:

   * Absolute neutrophil count (ANC) < 1,000/µL
   * Platelet count < 75,000/µL for subjects in whom < 50% of bone marrow nucleated cells are plasma cells; or a platelet count < 30,000/ µL for subjects in whom ≥ 50% of bone marrow nucleated cells are plasma cells
   * Creatinine Clearance < 45 mL/min according to Cockcroft-Gault formula
   * Corrected serum calcium > 14 mg/dL (> 3.5 mmol/L)
   * Hemoglobin < 8 g/dL (< 4.9 mmol/L; prior RBC transfusion or recombinant human erythropoietin use is permitted)
   * Serum glutamic oxaloacetic transaminase (SGOT)/ aspartate aminotransferase (AST) or Transaminase, serum glutamic pyruvic (SGPT)/ alanine aminotransferase (ALT) > 3.0 x upper limit of normal (ULN)
   * Serum total bilirubin > 1.5 x ULN
5. Subjects with prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years. Except the following: Basal cell carcinoma of the skin, Squamous cell carcinoma of the skin, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative.
6. Subjects with previous therapy with Pomalidomide
7. Subjects with hypersensitivity to thalidomide, lenalidomide, bortezomib, boron, mannitol, or dexamethasone
8. Subjects with ≥ Grade 3 rash during prior thalidomide or lenalidomide therapy
9. Subjects who had any of the following within the last 14 days of initiation of study treatment: Plasmapheresis, Major surgery (kyphoplasty is not considered major surgery), Radiation therapy, Any anti-myeloma drug therapy
10. Subjects who have received any investigational agents within 28 days or 5 half-lives (whichever is longer) of treatment
11. Pregnant or breastfeeding females
12. Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception.
13. Subjects with known Human immunodeficiency virus (HIV) positivity or active infectious hepatitis A, B, or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-02-15 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 2 years
  To determine the maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Adverse events | Up to 7 years
  Number of participants with adverse events (AEs)
Overall Survival | Up to 7 years
  Number of patients alive
Response Rate | Up to 7 years
  Overall response rate based on the International Myeloma Working Group (IMWG) Uniform response criteria
Duration of response | Up to 7 years
  Time from the initial documented response to confirmed disease progression
Time to response | Up to 7 years
  Time from enrollment to the first documented response

CONTACTS AND LOCATIONS:
Overall Officials: Amine Bensmaine, MD, Study Director — Celgene
Locations (6):
- United States (6):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Background] Richardson PG, Hofmeister CC, Raje NS, Siegel DS, Lonial S, Laubach J, Efebera YA, Vesole DH, Nooka AK, Rosenblatt J, Doss D, Zaki MH, Bensmaine A, Herring J, Li Y, Watkins L, Chen MS, Anderson KC. Pomalidomide, bortezomib and low-dose dexamethasone in lenalidomide-refractory and proteasome inhibitor-exposed myeloma. Leukemia. 2017 Dec;31(12):2695-2701. doi: 10.1038/leu.2017.173. Epub 2017 Jun 2. PMID 28642620
- [Background] Pelligra CG, Parikh K, Guo S, Chandler C, Mouro J, Abouzaid S, Ailawadhi S. Cost-effectiveness of Pomalidomide, Carfilzomib, and Daratumumab for the Treatment of Patients with Heavily Pretreated Relapsed-refractory Multiple Myeloma in the United States. Clin Ther. 2017 Oct;39(10):1986-2005.e5. doi: 10.1016/j.clinthera.2017.08.010. Epub 2017 Sep 28. PMID 28967482
- [Background] Moreau P, Dimopoulos MA, Richardson PG, Siegel DS, Cavo M, Corradini P, Weisel K, Delforge M, O'Gorman P, Song K, Chen C, Bahlis N, Oriol A, Hansson M, Kaiser M, Anttila P, Raymakers R, Joao C, Cook G, Sternas L, Biyukov T, Slaughter A, Hong K, Herring J, Yu X, Zaki M, San-Miguel J. Adverse event management in patients with relapsed and refractory multiple myeloma taking pomalidomide plus low-dose dexamethasone: A pooled analysis. Eur J Haematol. 2017 Sep;99(3):199-206. doi: 10.1111/ejh.12903. Epub 2017 Jun 14. PMID 28504846